CLINICAL TRIAL: NCT06417658
Title: A Comparison of Cosmetic Results in Terms of Scar Assessment and Complications in Endoscopic Supraorbital Eyebrow Craniotomy vs Conventional Craniotomy for Frontal Skull Base Lesions
Brief Title: Comparing Cosmetic Outcomes: Endoscopic vs. Conventional Craniotomy for Frontal Skull Base Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Syeda Ayesha Hashmi, Post Graduate Resident, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp122
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: The study employs a structured protocol involving random allocation to groups, preoperative assessments, surgery, postoperative follow-ups, and statistical analysis. It aims to evaluate differences in scar appearance, spread, erythema, suture marks, hypertrophy/atrophy, and overall impression between the two surgical approaches using the Scar Cosmesis Assessment Rating (SCAR) scale. Additionally, patient-reported outcomes such as itch and pain will be examined. This model ensures comprehensive evaluation of cosmetic outcomes and patient satisfaction, providing valuable insights to inform treatment regimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Supraorbital Eyebrow Craniotomy (Experimental): his minimally invasive neurosurgical procedure accesses brain tumors by making a small incision within the eyebrow, providing access to pathologies of the anterior skull base. Compared to traditional frontal craniotomy, this approach aims to minimize tissue disruption, potentially reducing postoperative complications and improving cosmetic outcomes. The procedure involves precise surgical techniques guided by endoscopic visualization, allowing for targeted tumor resection while preserving surrounding healthy tissue. Additionally, the use of smaller incisions may lead to reduced scarring and faster recovery times compared to conventional approaches.
  Interventions: Procedure: Endoscopic Supraorbital Eyebrow Craniotomy
- Conventional Frontal Craniotomy (Active Comparator): This arm represents the standard surgical approach for treating frontal skull base lesions. In this arm, surgeons perform the craniotomy through a conventional frontal approach rather than the endoscopic supraorbital eyebrow approach. This arm serves as the comparator against the experimental arm to evaluate the differences in cosmetic outcomes, scar assessment, and complications between the two surgical techniques.
  Interventions: Procedure: Conventional Frontal Craniotomy

INTERVENTIONS:
Procedure: Endoscopic Supraorbital Eyebrow Craniotomy — The Endoscopic Supraorbital Eyebrow Craniotomy is a minimally invasive neurosurgical procedure used to access and remove brain tumors located in the anterior skull base region. In this approach, surgeons make a small incision within the eyebrow area to gain access to the underlying pathology, avoiding larger incisions and more extensive tissue disruption associated with traditional open craniotomies.
  Arms: Endoscopic Supraorbital Eyebrow Craniotomy
Procedure: Conventional Frontal Craniotomy — The Conventional Frontal Craniotomy is a traditional surgical approach used to access and treat lesions located in the frontal region of the skull base. In this procedure, surgeons make a single or multiple large incisions in the scalp overlying the frontal bone to gain access to the underlying pathology.
  Arms: Conventional Frontal Craniotomy

SUMMARY:
This research study will compare the cosmetic outcomes, specifically scar assessment and complications, between two surgical approaches for treating frontal skull base lesions: the endoscopic supraorbital eyebrow craniotomy and the conventional frontal craniotomy. The study will aim to evaluate the differences in scar appearance, spread, erythema, suture marks, hypertrophy/atrophy, and overall impression between the two approaches using the Scar Cosmesis Assessment Rating (SCAR) scale. Additionally, it will examine patient-reported outcomes such as itch and pain. The study will follow a structured protocol, including random allocation to groups, preoperative assessments, surgery, postoperative follow-ups, and statistical analysis. It will emphasize the importance of understanding cosmetic outcomes to improve patient satisfaction and inform treatment regimens.

DETAILED DESCRIPTION:
The proposed research study will undertake a comparative analysis of the cosmetic outcomes associated with two distinct surgical approaches utilized in the treatment of frontal skull base lesions: the endoscopic supraorbital eyebrow craniotomy and the conventional frontal craniotomy. This investigation will primarily focus on evaluating scar assessment and complications arising from these surgical procedures.

1. Surgical Approaches: The study will compare two different techniques: the endoscopic supraorbital eyebrow craniotomy, which is a minimally invasive neurosurgical procedure involving a small incision within the eyebrow to access anterior skull base pathologies, and the conventional frontal craniotomy, a traditional approach involving a larger incision.
2. Purpose: The primary objective will be to assess and compare the cosmetic outcomes, particularly scar appearance and related complications, between these two surgical methods. The emphasis will lie on evaluating parameters such as scar spread, erythema, suture marks, hypertrophy/atrophy, and overall impression using the Scar Cosmesis Assessment Rating (SCAR) scale.
3. Study Protocol:

   Random Allocation: Patients will be randomly assigned to either the endoscopic supraorbital eyebrow craniotomy group or the conventional frontal craniotomy group.

   Preoperative Assessment: Comprehensive preoperative evaluations will be conducted to ascertain baseline data and ensure suitability for surgery.

   Surgery: Patients will undergo the assigned surgical procedure based on random allocation.

   Postoperative Follow-up: Close monitoring of patients post-surgery to assess scar healing and detect any complications.

   Data Collection: Data regarding scar assessment, complications, patient-reported outcomes, and other relevant parameters will be collected at specified intervals.

   Statistical Analysis: Rigorous statistical analysis of collected data will be conducted to draw comparisons and conclusions regarding cosmetic outcomes between the two surgical approaches.
4. Patient-Reported Outcomes: In addition to clinician-assessed scar parameters, the study will also consider patient-reported outcomes such as itch and pain, providing a comprehensive understanding of the patient experience following these surgical interventions.
5. Significance: The study will underscore the significance of evaluating cosmetic outcomes in neurosurgical procedures, aiming to enhance patient satisfaction and inform treatment decisions. By comparing the two surgical approaches, the research will seek to contribute valuable insights that may lead to the refinement of surgical techniques and improved patient care.

Overall, this proposed research endeavors to offer a detailed examination of the cosmetic results associated with endoscopic supraorbital eyebrow craniotomy versus conventional frontal craniotomy, thereby facilitating informed decision-making and optimizing patient outcomes in the management of frontal skull base lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having frontal skull base lesion on MRI
2. Lesion size <5cm on MRI with IV contrast
3. Both male and female
4. 25-65 years of age

Exclusion Criteria:

1. Patients with redo surgery (on medical record)
2. Lesion size >5cm
3. Vascular tumors
4. Previous trauma
5. Anticoagulant medications
6. Comorbidities(uncontrolled hypertension and diabetes)
7. Skin diseases

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Comparing Cosmetic Outcomes in Frontal Craniotomy Approaches | 12 months
  Comparison between two surgical approaches for treating frontal skull base lesions: the endoscopic supraorbital eyebrow craniotomy and the conventional frontal craniotomy will be made.
  The Scar Cosmesis and Assessment Rating (SCAR) scale will be used to determine the cosmetic outcome of the approach. The range of SCAR scale is 0 to 15. A score ≤ 5 on the SCAR scale will be considered cosmetic success. (Ziai et. al., 2022)

IPD SHARING:
Plan to Share IPD: No